CLINICAL TRIAL: NCT01520480
Title: Pathological Subtrochanteric Fractures in 194 Patients. A Comparison of Outcome After Surgical Treatment of Pathological and Non-pathological Fractures.
Brief Title: Pathological Subtrochanteric Fractures in 194 Patients
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Rudiger Weiss, Clinical professor, Karolinska University Hospital
Other Study IDs: 206/02
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Subtrochanteric Femur Fractures
Keywords: survival after surgery; Pathological Subtrochanteric Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-pathological fracture: Non pathological subtrochanteric femur fractures
- Pathological fracture: Pathological subtrochanteric fractures

SUMMARY:
In this study, the investigators analyze a consecutive series of patients operated for pathological subtrochanteric femur fracture to describe survival and reoperation rates after surgery and to identify risk factors for death. Moreover, the investigators include a cohort of patients with non-pathological subtrochanteric fractures for comparison.

DETAILED DESCRIPTION:
The Scandinavian Sarcoma Group (SSG) has initiated a Skeletal Metastasis Register in 1999. The Register is a quality-control database which prospectively collects individual-based information on patients operated for skeletal metastases in the long bones and pelvis. Data on patient identity, age, sex, primary tumor, location of metastases, type of pathological fracture, and perioperative treatment were gathered. Information concerning surgical procedures such as method of fixation, type of implant, and postoperative complications are registered. Moreover, some clinical data such as pain levels (no, light, moderate, strong, or severe pain), pain medication use, mobility, and the Karnofsky performance score are recorded.

We will identify all patients surgically treated for pathological subtrochanteric femur fractures during 1999-2009.

The Stockholm Hip Fracture Group provides data on the reference group. During 2003, a consecutive series of patients with acute non-pathological subtrochanteric femur fractures treated in Stockholm were included in a prospective cohort study. The regional ethical review board located at the Karolinska Institutet approved the study (DNR 206/02).

The aim of this study is to analyze survival and reoperation rates of patients operated for pathological subtrochanteric femur fracture. We want compare those findings with a cohort of patients with non-pathological subtrochanteric fractures.

ELIGIBILITY:
Inclusion Criteria:

* All patients with pathological subtrochanteric femur fractures register in the Scandinavian Sarcoma Group Register

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pathological subtrochanteric femur fractures.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 1999-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)